CLINICAL TRIAL: NCT03111238
Title: The Efficacy and Safety of Intra-arterial Administration of REX-001 to Treat Ischemic Rest Pain in Subjects With Critical Limb Ischemia (CLI) Rutherford Category 4 and Diabetes Mellitus (DM): a Pivotal, Placebo-controlled, Double-blind, Parallel-group, Adaptive Trial
Brief Title: The Efficacy and Safety of REX-001 to Treat Ischemic Rest Pain in Subjects With CLI Rutherford Category 4 and DM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped due to inactivity
Sponsor: Ixaka Ltd (Industry)
Collaborators: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REX-001-004
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Peripheral Arterial Disease (PAD); Diabetes Mellitus (DM); Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Cardiovascular Disease; Critical Limb Ischemia (CLI)
Keywords: Autologous; Bone Marrow-derived Mononuclear Cells (BM-MNCs); Advanced Therapy Medicinal Product (ATMP); Tissue-engineered Medicinal Product; Revascularization; Angiogenesis; Vasculogenesis; Arteriogenesis
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REX-001 (Experimental): REX-001 is a cell suspension of autologous BM-MNCs composed of several mature cell types.
  Interventions: Drug: REX-001
- Placebo (Placebo Comparator): The final formulation of the placebo will be a diluted suspension of red blood cells.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REX-001 — REX-001 is administered through an intra-arterial catheter.
  Arms: REX-001
Drug: Placebo — Placebo is administered through an intra-arterial catheter.
  Arms: Placebo

SUMMARY:
This trial is a pivotal, placebo-controlled, double-blind, parallel-group, adaptive trial conducted in subjects with DM and CLI Rutherford Category 4. Minimisation will be used to assign eligible subjects in a 2:1 ratio to receive a single intra-arterial administration of REX-001 or matching placebo into the index limb.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 to ≤ 85 years.
2. Diagnosis of Type I or II DM, established more than one year ago.
3. Glycosylated hemoglobin (HbA1c) < 9%.
4. Subjects with poor or no (surgical or endovascular) revascularization option classified as CLI Rutherford Category 4. The blood circulation in these subjects must be compromised at screening, defined as:

   * Ankle systolic pressure < 50 mm Hg, or
   * Toe systolic pressure < 30 mm Hg, or
   * TcpO2 < 30 mm Hg, and
   * Flat or barely pulsatile ankle or metatarsal PVR
5. In the opinion of the Investigator, the subject is controlled on medical therapy indicated for CLI (unless there is a documented contraindication or intolerance) and pain management is optimized.
6. Women of childbearing potential (i.e., fertile, following menarche and until becoming post-menopausal unless permanently sterile) must have a negative pregnancy test at screening. Men and women who are sexually active shall use effective contraceptive methods for the duration of their participation in this study if the partner of the male participant, or if the female participant is of childbearing potential.

Exclusion Criteria:

1. Advanced CLI defined as presence of major tissue loss as significant ulceration/gangrene proximal to the metatarsal heads (CLI Rutherford Category 6). Significant ulceration/gangrene means any ulceration that extends beyond the subcutaneous tissue layer, or any gangrene or tissue necrosis proximal to the metatarsal heads.
2. CLI Rutherford Category 5.
3. Uncontrolled or untreated proliferative retinopathy.
4. Failed surgical or endovascular revascularization on the index leg within 10 days after the procedure.
5. Subjects in whom arterial insufficiency in the lower extremity is the result of acute limb ischemia or an immunological or inflammatory or non-atherosclerotic disorder (e.g., thromboangiitis obliterans (Buerger's Disease), systemic sclerosis (both limited and diffuse forms).
6. Clinical evidence of invasive infection on index leg defined as major tissue loss at the mid-foot or heel involving tendon and/or bone, and/or when intravenous antibiotics are required to treat the infection according to the Investigator.
7. At screening, the presence of only neuropathic ulcers on the index leg.
8. Amputation at or above the talus on the index leg.
9. Planned major amputation within the first month after randomization.
10. On the index leg, use of concomitant wound treatments not currently approved for ischemic wound-healing within 30 days prior to screening or plans to initiate new, nonstandard-of-care treatments to the index leg during the trial.
11. Blood clotting disorder not caused by medication (e.g., thrombophilia).
12. Severe hypertension according to the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure.
13. A platelet count < 50,000/ μL.
14. International normalised ratio (INR) > 1.5. For patients on anticoagulant medication an INR > 1.5 is allowed, provided that the Investigator and the haematologist consider the patient eligible to collect BM.
15. Evidence of moderate to severe hepatocellular dysfunction according to the treating physician.
16. Positive test for human immunodeficiency virus 1 (HIV 1), HIV 2, hepatitis B virus (HBV), hepatitis C virus (HCV) or Treponema pallidum.
17. Subjects who may not be healthy enough to successfully complete all protocol requirements including BM collection, or who are not expected to survive more than 12 months, or in whom results may be particularly difficult to assess, as assessed by the Investigator.
18. Subjects who participate in another clinical interventional trial.
19. Subjects who have been treated with experimental medication within 30 days of screening.
20. Subjects who were treated with other cell therapies for CLI within the last 12 months preceding the screening visit.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Complete relief of ischemic rest pain without developing ischemic lesions on the index leg. | The primary endpoint for this trial will be assessed at 12 months.
  Change in Rutherford classification from CLI Category 4 to Category 3 or lower 12 months after administration of REX-001 or placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Wagener, MD, Study Director — Ixaka Limited
Locations (15):
- Czechia (2):
  - Fakultní nemocnice Ostrava, Ostrava
  - Vitkovicka nemocnice a. s. Vaskularni centrum, Ostrava
- Klinikum der Goethe-Universität Frankfurt, Frankfurt, Germany
- Pécsi Tudományegyetem, PTE-KK I. sz Belgyógyászati Klinika, Pécs, Hungary
- Instytut Hematologii i Transfuzjologii, Warsaw, Poland
- Centro Hospitalar de São João, Porto, Portugal
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - First site: Hospital Universitario Reina Sofía, Córdoba
  - Complejo Hospitalario Universitario de Granada, Hospital del Campus de la Salud, Granada
  - Hospital Universitario de la Princesa, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen de Valme, Seville

IPD SHARING:
Plan to Share IPD: Undecided